CLINICAL TRIAL: NCT02000063
Title: Long-term Outcomes Following Treatment of Recently Acquired Hepatitis C Virus Infection.
Brief Title: Australian Trial in Acute Hepatitis C Recall Study
Acronym: ATAHC Recall
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Other Study IDs: VHCRP1105; VHCRP1105 (Other: Kirby-VHCRP)
Record Dates: First submitted 2013-11-12; First posted 2013-12-03 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Acute Hepatitis C
Keywords: Hepatitis C; acute; early chronic
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored serum and peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No

SUMMARY:
A single long-term follow up assessment of an established multi-centre, prospective longitudinal cohort study of patients for clinical, psychosocial, immunovirological outcomes 4 to 8 years after previous treatment for recently acquired hepatitis C virus infection.

DETAILED DESCRIPTION:
The study aims are:

1. To evaluate the effect of successful prior treatment or spontaneous clearance of recently acquired HCV infection on long-term quality of life, social functioning, injecting behaviour, mental health and liver health.
2. To assess the incidence of HCV re-infection following prior treatment induced clearance or spontaneous clearance of recently acquired chronic HCV infection.
3. To determine predictors of HCV re-infection following recently acquired HCV infection treatment.
4. To determine frequency and predictors of new mixed and superinfections in ATAHC subjects with persistent viraemia.
5. To add to a tissue repository of serum and PBMCs from well-characterised patients treated for recently acquired HCV infection to allow future examination of the role of other variables that may potentially impact on the prognosis and outcomes of early HCV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrolment in the Australian Trial of Acute Hepatitis C Virus Infection (ATAHC) Study.
* Provision of written, informed consent.

Exclusion Criteria:

* In the opinion of the investigator that the patient is not able to provide informed consent.
* Inability or unwillingness to comply with study collection requirements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated 60 participants will be recruited from 3 study sites: St Vincent's Hospital, Sydney; The Alfred Hospital, Melbourne; Royal Adelaide Hospital, Adelaide.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Long-term effects of HCV clearance | 4 to 8 years from initial infection
  Health related quality of life (measured by SF-12) Social functioning (measured by OTI survey) Injecting behaviour Mental health (measured by DASS and MINI) Liver health (measured by FibroScan and biochemical markers)

SECONDARY OUTCOMES:
Incidence of HCV re-infection | 4 to 8 years from initial infection
  Rate of HCV RNA positivity in patients previously HCV RNA negative.

OTHER OUTCOMES:
Predictors of HCV re-infection | 4 to 8 years from initial infection
  Associations of HCV re-infection in those with HCV RNA positivity who were previously HCV RNA negative.
Incidence and predictors of HCV mixed and superinfections in those with persistent viraemia. | 4 to 8 years from initial infection
  Rate (or proportion over average years of follow-up) of new mixed HCV RNA infections in those with persistent viraemia and no prior evidence of multiple HCV infection.
Collection of specimens for future immunological or virological research. | 4 to 8 years from initial infection
  Stored serum and peripheral blood mononuclear cells.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MBChB, MRCP (UK), FRACP, PhD, Principal Investigator — University of New South Wales, Syndey Australia
Locations (3):
- Australia (3):
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria

REFERENCES:
- See also: UNSW Kirby Institute for infection and immunity in society Homepage — http://www.kirby.unsw.edu.au